CLINICAL TRIAL: NCT00496886
Title: Imaging the Cognitive Modulation of Pain
Brief Title: Determining How the Nervous System Processes Pain in Adults With Fibromyalgia
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01AR050969 (NIH); R01AR050969 (NIH); 1R01AR050969-01A1 (NIH)
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2013-02

CONDITIONS: Fibromyalgia; Rheumatoid Arthritis
Keywords: Pain; Nociception
MeSH Terms: conditions — Fibromyalgia; Arthritis, Rheumatoid; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Fibromyalgia (FM) is a disabling chronic disorder characterized by widespread muscle pain, fatigue, and multiple tender points, specific places on the body that become painful with only slight pressure. Pain associated with FM cannot be explained medically, often leading to a delayed diagnosis and delayed treatment. The purpose of this study is to evaluate how the nervous system, specifically the brain, processes pain in women with FM.

DETAILED DESCRIPTION:
The cause of FM remains unknown, and more than half of all FM patients do not experience adequate pain relief from current treatment. Identifying the mechanisms of unexplained pain in people with FM is necessary to develop more beneficial treatments. One possible cause of FM may be associated with problems in how the body processes pain. People with FM appear to be hypersensitive to stimuli that normally are not painful. Specifically, the brain and spinal cord may not signal sensations correctly, resulting in abnormal pain sensations. This study will use functional magnetic resonance imaging (fMRI) to examine how pain is processed in the brain of adults with FM compared with adults with rheumatoid arthritis (RA), another chronic disease characterized by long-term pain with a known cause. This study will also determine the effect that anticipation and attention have on the processing of nonpainful stimuli in women with FM and RA. Both groups of people will also be compared to a control group of healthy people.

Participants in this study will include only women. This study will include two study visits that will occur on separate days. Each study visit will last from 2 to 3 hours. During the first study visit, participants will complete questionnaires. They will then rate heat stimuli applied to their hand and perform mental tasks while in a mock MRI machine. The mental tasks will consist of naming the color of words. Some participants will receive nonpainful heat stimuli; others will receive both painful and nonpainful heat stimuli. During the second study visit, participants will undergo the exact same procedures while in an actual MRI machine. There will be no follow-up visits for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FM or RA OR healthy
* Right-handed

Exclusion Criteria:

* Diagnosis of depression
* Using illegal drugs
* Claustrophobic
* Metal objects in body
* Require cardiovascular, high-dose antidepressant, or certain analgesic medications

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community and primary care clinic samples.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2006-04; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Brain responses to pain | Single experimental session
  The study determines brain responses to pain in both healthy participants and those with fibromyalgia under conditions designed to manipulate anticipation and attention.

SECONDARY OUTCOMES:
Physical activity | one week
  The study measures physical activity the week prior to brain imaging
Brain white matter | single experimental session
  The study measures white matter using diffusion tensor imaging methods

CONTACTS AND LOCATIONS:
Overall Officials: Dane B. Cook, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States